CLINICAL TRIAL: NCT04747522
Title: SARS-CoV-2 Cellular and Humoral Immune Response Following Vaccination of Kidney Transplant Recipients and Healthy Controls
Brief Title: Severe Acute Respiratory Syndrome Corona Virus 2 (SARS-CoV-2) Immune Kidney Transplant Study (COVID-19)
Acronym: SCV-KTx-imm
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anders Åsberg, Head of Laboratory, Oslo University Hospital
Other Study IDs: 227626
Record Dates: First submitted 2021-02-04; First posted 2021-02-10 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Kidney Transplant Infection; SARS-CoV Infection
Keywords: Vaccination; Humoral; Cellular
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Serum Isolated blood cells DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Kidney Transplanted patients: Kidney transplanted patients transplanted at least 6 months prior to SARS-CoV-2 vaccination. Vaccination according to national plan with messenger Ribonucleic acid (mRNA) vaccine
  Interventions: Drug: SARS-CoV-2 vaccine
- Healthy controls: Healthy hospital staff receiving SARS-CoV-2 mRNA vaccine as being front line Healthcare workers.
  Interventions: Drug: SARS-CoV-2 vaccine

INTERVENTIONS:
Drug: SARS-CoV-2 vaccine — SARS-CoV-2 vaccines currently on market, i.e. Pfizer/BioNTech and Moderna

SUMMARY:
None of the vaccines approved, or in clinical trials, have so far been tested on transplanted patients. If they produce an immune response to the Spike protein of SARS-CoV-2 it is unknown how long the protective immunity will last.

Not all immune responses are equal. The investigators will quantify immune cell subsets with flow and mass cytometry analyses to describe the phenotype of responding immune cells, including specific T cells. If not already established, patient human Leukocyte antigen (HLA) genotypes will be typed.

In order to compare the immune responses with healthy individuals a control group of hospital employees will be included and sampled before and after vaccination according to the same time schedules as the kidney transplanted patients.

DETAILED DESCRIPTION:
Kidney transplanted patients with post-transplant follow-up visits at the national transplant center in Norway will be included before they are SARS-CoV-2 vaccinated. As a control group the investigators will include blood samples from healthy volunteers (hospital employees) that receive vaccine as first line health care workers.

Baseline blood samples will be obtained before vaccination. The vaccination will be performed according to the national procedures and not necessarily by the hospital. Following vaccination, all patients and controls will have blood drawn 7-10 days as well as 4-6 weeks after the second dose. Depending on the results of the immunity testing the patients and controls may be invited to additional blood sampling up or at specific time points to two years following vaccination.

At each blood sampling and at the time of both vaccinations the systemic exposure of tacrolimus will be assessed in kidney transplanted patients.

All samples will be analyzed with validated assays for SARS-CoV-2 immunoglobulin G (IgG) (anti-receptor binding domain (RBD) spike protein) using ELISA, flow cytometry bead arrays and SARS-CoV-2 neutralization assays or comparable techniques. Cells will be analyzed by flow and mass cytometry for activation and phenotype markers, and with functional assays for responsiveness (e.g. proliferation and cytokine production). Samples will be HLA-typed if HLA-genotype if not already established.

ELIGIBILITY:
Inclusion Criteria:

* Patients transplanted with a kidney (only) at least 6 months before vaccination OR healthy volunteer first line health care workers at OUS.
* Age of 18 years or older (also for controls).
* Standard immunological risk at transplantation (i.e. no donor specific HLA antibodies (DSA)) and not performed an ABO blood-type-incompatible transplantation.
* No treatment for rejection episodes the last 6 months before inclusion.
* Immunosuppressive therapy including tacrolimus, mycophenolate and prednisolone.
* Stable graft-function the last 6 months.
* S-creatinine < 200 μmol/L (also for controls).
* Signed informed consent to participate in the study (also for controls).

Exclusion Criteria:

* Three or more previous transplantations.
* Hemoglobin level below 10 g/dL (also for control).
* Leukopenia defined as total lymphocyte count < 2 X 109 (also for controls).
* Previous treatment with anti-thymocyte antibodies (ATG) or rituximab.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult, standard risk kidney transplanted patients on tacrolimus based immunosuppressive therapy are eligible for inclusion in the project.
  Adult, healthy Oslo university hospital (OUS) employees that receive vaccine as first line health care workers and that are not treated for any disease known to be a risk factor for severe COVID-19. These will be invited to participate via study information posted in the relevant clinics.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cellular immunological response | 1.5 months
  IgG antibodies against SARS-CoV-2 spike protein above assay limit of positive sample.
Humoral immunological response | 1.5 months
  T-cell reactivity against SARS-CoV-2 spike protein, including known mutation in the spike protein.

SECONDARY OUTCOMES:
Vaccine related side effects | 6 months
  Adverse drug reactions that have a reasonable relation to the vaccination, as assessed by the investigator

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Potential sharing of de-identified immunological data. Need specific ethical Committee approval for sharing